CLINICAL TRIAL: NCT02710032
Title: TransPrEP: Social Network-Based PrEP Adherence for Transgender Women in Peru
Acronym: TransPrEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: The Fenway Institute (Other); Brown University (Other); Asociación Civil Impacta Salud y Educación, Peru (Other)
Responsible Party: Principal Investigator, Jesse Clark, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R34MH104072 (NIH)
Record Dates: First submitted 2016-03-08; First posted 2016-03-16 (Estimated); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: HIV Infection
Keywords: Transgender women; HIV Pre-Exposure Prophylaxis; Adherence; Peru; Social Networks
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Social Network-Based Adherence Intervention
  Interventions: Behavioral: Social Network-Based Adherence Intervention; Behavioral: Social Media Platform
- Control (No Intervention): Control

INTERVENTIONS:
Behavioral: Social Network-Based Adherence Intervention — Participants in clusters randomized to the intervention arm will be asked to attend a series of weekly group workshops emphasizing a collective approach to HIV prevention and mutual support for PrEP adherence.
  Arms: Intervention
Behavioral: Social Media Platform — ii) Social Media Platform: The social media component of the intervention will include structured internet platforms designed to educate, motivate, and promote discussions of PrEP adherence within the participant network, unstructured participant-generated interactions to articulate and reinforce newly developed social norms within the network, and practical tools to support daily PrEP adherence.
  Arms: Intervention

SUMMARY:
The investigators propose a social network-based PrEP adherence intervention as part of a comprehensive, context-specific approach to HIV prevention for TW in Lima, Peru. In order to be effective, PrEP-based prevention strategies need to address not only biological efficacy, but also individual behavioral decision-making processes, interpersonal partnership contexts of risk, peer norms of sexual behavior and PrEP adherence, and structural access to prevention technologies. Using a health promotion behavioral model that combines Social Action Theory with social network theories of information dissemination and collective behavior change, the investigators propose to develop and refine a network-based intervention that promotes PrEP adherence in the existing social networks of TW. Formative research will outline individual, partner-level, and network-based contexts of sexual risk behavior, patterns of social network interactions, anticipated adoption and use of new prevention technologies, and optimal content for a PrEP adherence intervention. Findings will be used to define the elements of a prevention intervention using social networks of TW and social media technologies to generate, implement, and reinforce social norms of PrEP adherence and risk behavior reduction for TW.

DETAILED DESCRIPTION:
Pre-Exposure Prophylaxis (PrEP) has biological efficacy in reducing risk for HIV acquisition but its clinical effectiveness is strongly influenced by patient adherence, which is in turn influenced by social and behavioral factors. Trials conducted among serodiscordant heterosexual African couples who were engaged in supportive romantic partnerships found PrEP to be highly effective for HIV prevention. In contrast, studies with socially marginalized populations in Latin America without strong interpersonal support networks, such as transgender women (TW), found substantially lower levels of adherence and, as a result, effectiveness. We believe that new, social network-based strategies to promote PrEP adherence, coupled with behavioral interventions to minimize risk compensation, will be critical to controlling the spread of HIV among TW in Latin America.

TW in Peru are at high risk for HIV infection (30-33% HIV prevalence) and in urgent need of new approaches to prevention that adequately address HIV risk as part of their life contexts. Due to their social and economic marginalization and lack of support from traditional neighborhood and family networks, TW frequently neglect traditional approaches to HIV/STI prevention that have been developed for men who have sex with men (MSM), and report high rates of compensated sex, unprotected intercourse, and sexually transmitted infection (STI) co-infections. Despite their socially marginalized status, communities of TW in Lima are frequently connected through dense social and geographic networks that provide support outside of traditional community systems, disseminate new information and ideas, and define and maintain standards of behavior. While these social networks provide a critical framework for the dissemination and maintenance of TW community norms, they have not previously been used as a framework for HIV prevention.

We propose a social network-based PrEP adherence intervention as part of a comprehensive, context-specific approach to HIV prevention for TW in Lima, Peru. In order to be effective, PrEP-based prevention strategies need to address not only biological efficacy, but also individual behavioral decision-making processes, interpersonal partnership contexts of risk, peer norms of sexual behavior and PrEP adherence, and structural access to prevention technologies. Using a health promotion behavioral model that combines Social Action Theory with social network theories of information dissemination and collective behavior change, we propose to develop and refine a network-based intervention that promotes PrEP adherence in the existing social networks of TW. Formative research will outline individual, partner-level, and network-based contexts of sexual risk behavior, patterns of social network interactions, anticipated adoption and use of new prevention technologies, and optimal content for a PrEP adherence intervention. Findings will be used to define the elements of a prevention intervention using social networks of TW and social media technologies to generate, implement, and reinforce social norms of PrEP adherence and risk behavior reduction for TW.

Aim 1. To conduct an open evaluation of a social network-based PrEP adherence intervention for TW in Peru. The intervention will be piloted with a group of 10-15 TW recruited from a social network within a single geographic area. Using a dynamic process of implementation, refinement, and re-implementation over a 6-month period, we will assess acceptability and feasibility of specific intervention and evaluation components. Data will be used to finalize the study design, intervention manual, and quantitative assessment tools for the pilot randomized controlled trial.

Aim 2. To conduct a pilot RCT of a social network-based PrEP adherence intervention for TW in Peru. The investigators plan to enroll 6 social network clusters of TW (3 clusters per arm, recruited from 2 seeds matched from 3 geographical areas in Lima, Peru) (total N=90 TW enrolled [15 TW per cluster] to achieve at least N=60 TW completers [10 TW per cluster]) that will be randomized to participate in either the network-based PrEP adherence intervention or a control intervention. The primary outcome will be adherence to PrEP (measured via laboratory analysis of presence of detectable drug in serum, laboratory analysis of presence of detectable drug in hair, and participant self-report). The major secondary outcome will be behavioral risk compensation, specifically the degree to which participants in the two arms do or do not modify HIV risk behaviors while taking PrEP. Behavioral and biological assessments will be conducted at Baseline, 3-month, and 6-month intervals.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older;
2. Identify as male-to-female transgender (e.g., "trans," "transgender," "travesti");
3. Report behavioral risk for HIV infection (UAI with at least one HIV-infected or unknown serostatus partner in the preceding 6 months);
4. HIV-uninfected by rapid test.

Exclusion Criteria:

1. Unable to provide informed consent, including people with severe mental illness requiring immediate treatment or with mental illness limiting their ability to participate (e.g., dementia);
2. HIV infection (Rapid HIV assay positive);
3. Active Hepatitis B infection (Hepatitis B Surface Antigen positive);
4. Renal insufficiency (Creatinine Clearance <50).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Serum Drug Level | 6 Months
  Serum monitoring of Truvada drug level

SECONDARY OUTCOMES:
Self-reported Adherence | 6 Months
  Self-reported adherence to Truvada
Hair Sample Drug Level | 6 Months
  Hair sample monitoring of Truvada drug level

CONTACTS AND LOCATIONS:
Overall Officials: Jesse L Clark, MD, MSc, Principal Investigator — UCLA Geffen School of Medicine
Locations (1):
- Asociacion Civil Impacta Salud y Educacion, Lima, Peru

IPD SHARING:
Plan to Share IPD: No
Due to restrictions on sharing of human subjects data, other researchers' requests for access to data will be reviewed and subject to approval by the relevant IRBs.